CLINICAL TRIAL: NCT02174016
Title: The Ketogenic Diet for Pediatric Acute Brain Injury
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Joyce Matsumoto, Health Sciences Assistant Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-001156A
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Brain Injuries
Keywords: Intensive Care Units; Pediatric
MeSH Terms: conditions — Brain Injuries | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Open label use of ketogenic diet in children with acute brain injury
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketogenic diet (Experimental): All subjects will be started on ketogenic diet formula feeding after enrollment for 2 weeks.
  Interventions: Dietary Supplement: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet

SUMMARY:
This is a prospective pilot study evaluating the safety and feasibility of implementing the ketogenic diet in children admitted to the pediatric intensive care unit with acute brain injury such as stroke, traumatic brain injury, and intracerebral hemorrhage. Animal studies suggest that in the aftermath of injury the brain's ability to use glucose as a fuel is impaired. The ketogenic diet is a high fat, low carbohydrate diet which is already used in clinical practice for the treatment of medication resistant epilepsy and is intended to switch the body over to burning fat rather than carbohydrates for fuel. In lieu of their standard tube-feeds, 5-10 children admitted to the PICU with these diagnoses will receive low carbohydrate, high fat ketogenic feeds for 2 weeks. We hypothesize that ketones will be detectable through serum tests and MRI spectroscopy studies of the brain within several days of diet initiation, and that there will be a low incidence of side effects and adverse events,

Measures of interest will include the incidence of kidney stones, excessive acidosis and excessive hypoglycemia. The feasibility of implementing this protocol for a larger efficacy trial will be assessed through serial measurements of blood glucose, beta-hydroxybutyrate (a type of ketone body), and serum bicarbonate levels. In addition, levels of ketone bodies within the brain will be measured through MRI spectroscopy sequence which will be acquired at the same time as a follow-up MRI brain study ordered for clinical purposes.

ELIGIBILITY:
Inclusion Criteria: children age -17 years admitted to the pediatric intensive care unit with acute brain injury such as acute stroke, severe traumatic brain injury, and intracerebral hemorrhage

Exclusion Criteria:

1. True milk allergy (anaphylaxis or severe rash)
2. Significant gastrointestinal injury precluding enteral feeding
3. Hepatic or renal insufficiency
4. History of nephrolithiasis
5. Severe acidosis (serum bicarbonate ≤ 17 mEq/L) resistant to correction
6. History of inborn error of metabolism
7. Preexisting epilepsy or developmental delay

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-06 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Increase in Beta-hydroxybutyrate level | 2 weeks
  Serum beta hydroxybutyrate levels will be checked daily, in order to determine how many days it will take to achieve elevated levels.

SECONDARY OUTCOMES:
Number of episodes of low blood glucose levels | 2 weeks
Number of episodes of low serum bicarbonate levels | 2 weeks
  Bicarbonate levels are expected to decrease because ketone bodies are acidic in nature, but episodes of excessively low bicarbonate levels will be assessed.
Number of subjects with MRI brain spectroscopy peaks corresponding to ketone body compounds, | 5 days
Number of subjects who develop kidney stones | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States